CLINICAL TRIAL: NCT01181999
Title: Phase II Trial of Rituximab (R) Augmentation Following R-CHOP (Cyclophosphamide, Doxorubicin, Vincristine, and Prednisolone) Induction Chemotherapy in Extremely Elderly Patients With Diffuse Large B Cell Lymphoma (DLBCL)
Brief Title: Rituximab Augmentation Following R-CHOP Induction Chemotherapy in Extremely Elderly Patients With Diffuse Large B Cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chonnam National University Hospital (Other)
Collaborators: Samsung Medical Center (Other); Asan Medical Center (Other); Severance Hospital (Other)
Responsible Party: Principal Investigator, Deok-Hwan Yang, Professor, Chonnam National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML25393
Record Dates: First submitted 2010-08-11; First posted 2010-08-16 (Estimated); Last update posted 2011-09-22 (Estimated); Status verified 2010-07

CONDITIONS: Lymphoma, Large B-cell, Diffuse
Keywords: diffuse large B-cell lymphoma; elderly patients; rituximab augmentation
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- rituximab (Experimental)
  Interventions: Drug: rituximab

INTERVENTIONS:
Drug: rituximab — A dose of 375mg/m2 rituximab will be administered intravenously on day 1 of first to fourth R-CHOP chemotherapy and on day 1, 8, 15, 22 of each augmentation chemotherapy.

SUMMARY:
Rituximab (R) plus CHOP (cyclophosphamide, doxorubicin, vincristine, and prednisolone) combination is considered as the new gold standard for the first-line treatment of elderly patients with diffuse large B-cell lymphoma (DLBCL).

The study is aimed to evaluate the overall response rate and the safety of four cycles of R-CHOP chemotherapy and followed by rituximab augmentation (weekly four times infusion) in newly diagnosed DLBCL patients with aged more than 70 years.

DETAILED DESCRIPTION:
1. Four cycles of R-CHOP chemotherapy for the induction treatment [Dose intensity of CHOP chemotherapy is modulated according to Charlson Comorbidity Index (CCI)]

   If patients with CCI <1
   * Rituximab: 375 mg/m2, day 1 every 3 weeks.
   * Conventional dose of CHOP chemotherapy repeat every 3 weeks.

   If patients with CCI ≥1
   * Rituximab: 375 mg/m2, day 1 every 3 weeks.
   * 75% of conventional CHOP repeat every 3 weeks.
2. Rituximab augmentation

   * Rituximab: 375 mg/m2, every week x 4 times.
   * Trimethoprim-sulfamethoxazole 1 tablet per day during augmentation

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed CD20 positive DLBCL
2. Age ≥ 70
3. Ann Arbor stage II, III and IV
4. No prior chemotherapy or radiotherapy for DLBCL
5. Performance status (Eastern Cooperative Oncology Group) ≤ 2
6. At least one or more bidimensionally measurable lesion(s)

   * ≥ 2 cm by conventional computerized tomography (CT)
   * ≥ 1 cm by spiral CT
   * skin lesion (photographs should be taken) ≥ 2 cm
   * measurable lesion by physical examination ≥ 2 cm
7. Cardiac ejection fraction ≥ 50% as measured by echocardiogram without clinically significant abnormalities
8. Adequate renal function: serum creatinine level < 2 mg/dL (177 μmol/L)
9. Adequate liver functions:
10. Adequate bone marrow functions:

    hemoglobin ≥ 9 g/dL absolute neutrophil count ≥ 1,500/μL and platelet count ≥ 75,000/μL, unless abnormalities are due to bone marrow involvement by lymphoma
11. Life expectancy more than 6 months
12. Informed consent

Exclusion Criteria:

1. Other subtypes of non-Hodgkin's lymphoma
2. Patients who transformed follicular lymphoma or other indolent lymphoma
3. Primary Central Nervous System (CNS) DLBCL
4. CNS involvement by lymphoma or any evidence of spinal cord compression.
5. Patients with a known history of human immunodeficiency virus (HIV) seropositivity or hepatitis C virus (+).
6. Any other malignancies within the past 5 years except curatively treated non-melanoma skin cancer or in situ carcinoma of cervix uteri
7. Pregnant or lactating women, women of childbearing potential not employing adequate contraception
8. Other serious illness or medical conditions

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-08; Primary Completion 2012-03 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
the overall response rate | three years after the completion of rituximab augmentation
  To evaluate the objective overall response rate of four cycles of R-CHOP and followed by four times weekly rituximab augmentation in exteremely elderly patients with DLBCL.
Number of patients with adverse events | three years
  All patients will be evaluated for the toxicity during the treatment. Toxicity is graded according to the National Cancer Institute Common Toxicity Criteria (NCI-CTC v3.0).

SECONDARY OUTCOMES:
progression-free survival | Three years after the completion of rituximab augmentation

CONTACTS AND LOCATIONS:
Locations (1):
- Chonnam National University Hwasun Hosptial, Jeollanam-do, South Korea